CLINICAL TRIAL: NCT07112118
Title: Multimodal Identification of Depressive Symptoms
Brief Title: Multimodal Identification of Depressive Symptoms in the Elderly
Acronym: multimodal
Status: Not yet recruiting | Type: Observational
Sponsor: Wuhan Mental Health Centre (Other)
Responsible Party: Sponsor
Other Study IDs: KY2025.0115.01; 72404094 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2025-07-17; First posted 2025-08-08 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Depression
Keywords: depression symptoms
MeSH Terms: conditions — Depression | interventions — Data Collection

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- non-depression: Elderly people without depressive symptoms
  Interventions: Other: data collection
- depression: Elderly people at risk of depression
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — Collect the facial expressions, audio, text and postural behavior data of the respondents using electronic devices.

SUMMARY:
Screening with depression scales alone is subjective, and relying on single-modal data often leads to incomplete identification of symptoms that are easily missed or misdiagnosed. In this study, we first aim to use artificial intelligence to construct a depression symptom recognition model, concatenate multimodal features such as facial expression, audio, text, and postural behavior, and deeply fuse them to construct a multimodal model.

ELIGIBILITY:
Inclusion Criteria:

* Elderly individuals aged 60 years or older.
* Residents of the community (with residence time of more than 6 months).
* Possessing certain reading, writing and comprehension skills, being able to communicate with researchers without obstacles, and being able to independently complete the measurement of various indicators or, although unable to independently fill out the questionnaire, being able to independently make evaluations of the questionnaire items.
* Those who have given informed consent.

Exclusion Criteria:

* Those who meet the diagnostic criteria for cognitive impairment (dementia) as stipulated in DSM-5, and/or who suffer from severe physical diseases (such as advanced cancer, cardiovascular and cerebrovascular diseases, etc.).
* Those who are undergoing antidepressant treatment.
* Elderly individuals who have had suicidal thoughts in any psychological assessment, should be referred to the psychological hotline platform in Wuhan.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly individuals aged 60 years or older
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Use the PHQ-9 (Patient Health Questionnaire - 9 ) to assess whether the respondents have depressive symptoms. The scale score is one point for each item. | 2025.09.01-2026.09.01
  If the PHQ-9 score is 5 or higher, it is determined as a positive sign of depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxv Yin, PhD, Study Chair — Huazhong University of Science and Technology
Locations (1):
- Wuhan Mental Health Center, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No